CLINICAL TRIAL: NCT05087082
Title: Early Transfer of Hospitalized Patients Including COVID-19 Patients to a Virtual Hospital at Home(vHaH)Model -a Clinical Feasibility Study.
Brief Title: Early Transfer of Hospitalized Patients Incl. COVID-19 to a Virtual Hospital at Home Model - a Clinical Feasibility Study
Acronym: Influenz-er
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nordsjaellands Hospital (Other)
Collaborators: Innovation Fund Denmark (Individual); University of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H-21014302
Record Dates: First submitted 2021-08-18; First posted 2021-10-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-06

CONDITIONS: Telemedicine; Epidemic Disease

STUDY DESIGN:
Intervention Model Description: The study is a clinical feasibility study. We anticipate to enroll 20 participants. Participants are admitted patients with a lower respiratory infection are 18 years of age or older and have been admitted at the hospital for at least 24 hour. additionally they must be and are considered suitable for home admission according o the inclusion- and exclusion criteria. The participants will be a part of the study until discharge or withdrawal of consent. If a next-of-kin is identified as primary informal caregiver this person is offered to take participate in the study as well. Follow-up questionnaires will be sent to all participants, and follow-up interviews will be performed after discharge.
Masking Description: Masking of participants is not possible due to the nature of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- App and Case Management system with algorithms (Other): Feasibility study of hospital at home model including telemedicine and specifically developed app and case management system
  Interventions: Other: Virtual Hospital at Home - Home admission of epidemic patients

INTERVENTIONS:
Other: Virtual Hospital at Home - Home admission of epidemic patients — Admitting COVID-19 patients at home

SUMMARY:
This study will be part of a larger, 'virtual hospital-at-home' (vHaH) project called Influenz-er. vHaH is a care model designed to deliver medical care in the home, as a substitute for a continued inpatient hospital admission. This study will be a clinical feasibility study, which will be used to guide the framing and design of the final telemedicine supported vHaH model for hospitalized patients.

DETAILED DESCRIPTION:
This study will be part of a larger, 'virtual hospital-at-home' (vHaH) project called Influenz-er. vHaH is a care model designed to deliver medical care in the home, as a substitute for a continued inpatient hospital admission. An underlying rationale for the development of vHaH is that, by avoiding the hospital environment, fragile and older persons may experience high-quality care that is associated with fewer complications, and higher treatment satisfaction for patients and their families. Various versions of home-hospital models have been implemented during the COVID-19 pandemic crisis, but in many situations out of need and so far, only very limited documented experience from sound research approaches is available in the medical literature. This study will be a clinical feasibility study, which will be used to guide the framing and design of the final telemedicine supported vHaH model for hospitalized patients including epidemic patients. We apply our experience from 5 months of clinical small scale testing (Sept 2021 - Jan 2022) of the light version of the final vHaH model on hospitalized patients (the technology and workflows of the vHaH model were tested by in-patients under their hospital stay) to implement this novel model in the safest possible way. The vHaH model will be offered exclusively to moderately ill (not severely ill) patients with respiratory infections including COVID-19.

The overall aim of Influenz-er, is to develop and implement a novel telemedicine monitoring and communication model, that will enable safe admission of epidemic patients in their homes. We will implement this novel model in the safest possible way, and initially offer the vHaH model to patients conventionally admitted with COVID-19 illness or other lower respiratory tract infections causing pneumonia. Conversion to vHaH admission will be effectuated after an assessment by a medical infectious disease specialist if the patient is assessed to be ready to continue the hospital admission safely from home, under continued monitoring and treatment responsibility by the hospital.

Based on a Cochrane review this innovative alternative to conventional hospitalization, is expected to benefit patients who will remain in the comfort of their own homes. This model could potentially increase patient and next of kin quality of life and treatment satisfaction, decrease risks of nosocomial complications and increase availability of emotional support from next of kin.

A hospital based Virtual Epidemic Center (VEC) is the center of the project, from where medical staff will monitor and communicate with patients admitted at home. Vital parameters and patient reported outcomes will be collected using a smart phone/tablet-based app. All data will be collected and processed in an algorithm to predict the impact of changes on disease severity. Algorithm and direct patient data will be displayed in real-time at the hospital in the VEC, allowing medical staff to continuously monitor their patients. In addition, daily virtual ward rounds conducted by staff in the VEC and when relevant by medical doctors (MD) from specialties of relevance to the patients' illness(es) will ensure close communication and relevant clinical assessments. A mobile medical team consisting of nurses and medical doctors (MD), will perform in-person patient evaluations, administer medication and perform other required daytime routine medical tasks.

The Influenz-er project governance structure consists of a Steering Committee with representation by the project partners Nordsjællands Hospital, University of Southern Denmark and Innovation Fund Denmark, an international Advisory Board and a national Consulting Group. Head of Clinical Research at Nordsjællands Hospital, Professor Thea Kølsen Fischer is principle investigator and project manager. The project team includes clinical experts with expertise within management of COVID-19 as well as health economic senior experts, PhD students, administrative research and innovation coordinators and health tech developers.

The objective of this feasibility study is to investigate and analyze relevant factors for admitting adult patients with LTRI including COVID-19 in a vHaH model to ascertain the likelihood of completing the vHaH model successfully.

Enrolment: Potential study patients will be identified by the general healthcare staff of the hospital COVID-19 ward, after a minimum of 24 hours of observation and conventional care, in order to ensure that the patients are in a stable phase of the disease. The healthcare staff of the hospital COVID-19 ward will be trained in, and instructed to, recognize potential eligible patients and subsequently inform the attending study personnel in the VEC. Study personnel will then assess the patients in the ward. The patients will receive oral and written information regarding the study and will be asked if they can identify a next of kin as a primary informal caregiver. Primary informal caregivers can be anyone and does not necessarily have to live with the patients or be the person who spends most time with the patients. The patients are not required to identify a primary informal caregiver in order to participate in the study. Patients with children in their household are not necessarily excluded, as the guidelines mention how to accommodate kids in the household. Current guidelines regarding self-isolation of SARS-CoV-2 positive individuals given by the Danish government will be applicable for patients admitted at home and their primary informal caregivers.

If the patients do identify a primary informal caregiver this person will be contacted and the oral and written information regarding the study, will be repeated for the identified primary informal caregivers. Study consent is obtained electronically via REDCap from patients and primary informal caregivers (if any) who are still interested in participating after having received information regarding the study. This is followed by the generation of an inclusion-ID for each via REDCap. To ensure that identified primary informal caregivers are taken into consideration, it is a requirement that both patients and primary informal caregivers agree to participate in the study. The study patients must accept that primary informal caregivers have the rights to terminate the HaH-admission and demand the conversion of the HaH-admission to a conventional hospital admission at any time. If potential study patients do not accept this term it will be considered as an exclusion criterion and the patients will not be considered eligible for the study.

Subsequently, the patients will be formally assessed for inclusion, in accordance with inclusion- and exclusion criteria. Included patients and primary informal caregivers (if any) will get a formal study-ID each. Study patients will receive and install the study app on a compatible device and the study personnel will ensure that study patients are educated in the basic functionality of the app.

Patients who do not meet the inclusion criteria will be either permanently or temporarily excluded and will retain their inclusion-ID. Age, gender and the reason of exclusion will be noted.

The first set of biometric data will be obtained within the hospital, assisted by the staff in order to secure the proper usage of the equipment. Furthermore, study patients will be equipped with a direct phone number for the VEC, which they can use to contact the personnel in the VEC independently from the app. All study patients are instructed to contact 112 in the case of a medical emergency requiring immediate medical assistance.

The study patients will be instructed to measure and upload biometrical data (body temperature, blood pressure, heart rate, respiratory frequency, oxygen saturation, blood glucose) at a frequency specified by the attending Medical Doctor (MD) in accordance with medical assessment, according to standard hospital early warning score (EWS)-screening. Furthermore, patients will be instructed to complete and upload the self-assessment questionnaire along with all biometric uploads using the app. Study patients with controlled comorbidities will be monitored and treated as per usual according to local applicable guidelines, and medical specialists will be available for collegial sparring as is the case during a conventional hospitalization.

The app will notify the study patients when it is time to upload a new set of biometrical and self-assessed data and notify upcoming planned virtual ward rounds. Adjustments to surveillance level will be communicated directly to study patients by attending personnel in the VEC.

After all relevant information has been confidently delivered and the patient has demonstrated capability to use the app correctly the study patients will be admitted at home by the VEC MD on duty. All study patients will be offered a free transfer home. If the study patients are still dependent on supplemental oxygen this will be installed in their home prior to the home admission, and the patients and their relatives will receive thorough instructions in how to use the oxygen equipment as well as how to behave with oxygen equipment at home.

ELIGIBILITY:
Inclusion Criteria for patients:

* Age ≥ 18 years of age
* Signed informed written and oral consent
* Lower tract respiratory infections, including contagious infection (e.g. SARS CoV 2 and Influenza).
* Considered not ready for discharge for at least 24 hours, assessed by attending MD in the COVID-19 ward.
* Patients are self-reliant or receives sufficient formal care to be care-independent of primary informal caregiver
* - Medically eligible for vHaH, including but not solely dependent of following conditions, assessed by the attending VEC MD:
* Actual condition assessed to be clinically stable.
* Green or yellow-tag triage based on vital parameters, including total adjusted EWS-score ≤6 and no adjusted single parameter score of 3 or above (See appendix 1)
* Requires less than 5L/min of oxygen supplement
* Stable or decreasing need for oxygen supplement
* Stable or decreasing paraclinical infection parameters such as C-reactive protein (CRP) etc.
* Home-based admission will be located within catchment area of the hospital (according to the official address of the individual).

Exclusion criteria

* Patients who cannot participate in interaction via App
* Lack of sufficient Danish language skills to understand and interact with requirements and staff at a patient safe level
* Patient residency cannot offer isolated room (COVID-19 patients only)
* Pregnancy

Inclusion criteria specific for primary informal caregivers (if any)

* Signed informed written and oral consent
* Study patient is included in the study
* Age ≥ 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-04-20 (Actual); Primary Completion 2023-09-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Percentage of all planned daily video supported ward rounds provided | through study completion, approximately 18 months
  successful protocol adherence is defined by 80%
Percentage of all planned self-measurements transmitted by patient | through study completion, approximately 18 months
  successful protocol adherence is defined by 80%
Percentage of all acute contact requests from patients handled within pre-defined time | through study completion, approximately 18 months
  successful protocol adherence is defined by 80%
Percentage of all non-acute contact requests from patients handled within pre-defined time | through study completion, approximately 18 months
  successful protocol adherence is defined by 80%
Percentage of all red alarms triggered by EWS-change handled within pre-defined time | through study completion, approximately 18 months
  successful protocol adherence is defined by 80%
Percentage of all yellow alarms triggered by EWS-change handled within pre-defined time | through study completion, approximately 18 months
  successful protocol adherence is defined by 80%
Number of recruited participants | through study completion, approximately 18 months
  recruitment success is defined as 80%
Number of drop-out participants | through study completion, approximately 18 months
  success is defined by brop out less than 10%
Number and type of outcome assessment completed by participants. | through study completion, approximately 18 months

SECONDARY OUTCOMES:
Patient related endpoints: Compound of clinical events | 30 days efter the discharge.
  Compound of clinical events:
  * Health care associated infections during home-based admission
  * Delirium during home-based admission
  * Thromboembolic events during home-based admission
  * Admittance to intensive care unit (ICU) during home-based admission
  * Respirator treatment following home-based admission
  * Intravenous antibiotic treatment during home-based admission
  * Intravenous antiviral treatment during home-based admission
  * Thirty-day readmittance rate post discharge
  * Mortality (associated, 7 days and 30 days)
Patient related endpoints: Loss of function | Three months after discharge
  SF-36
Patient related endpoints: Productivity losses | Three months after discharge of patient
  Number of days patient is absent from work during the period of sickness in relation to the admission, number of days patient is not able to perform daily tasks such as cooking, grocery shopping and house cleaning during the period of sickness in relation to the admission and number of days in isolation during the period of sickness in relation to the admission
Patient related endpoints: Self-perceived quality of care | Three months after discharge of patient
  Questionnaire 5
Next of kin related endpoints: Quality of Life | Three months after discharge of patient
  SF-36 (Questionnaire 3)
Next of kin related endpoints: Quality of Life | Three months after discharge of patient
  EQ-5D-5L
Next of kin related endpoints: Caregiver strain | Two weeks after discharge of the patient
  Zarit Burden Interview (Questionnaire 6)
Next of kin related endpoints: Productivity losses | Three months after discharge of patient
  Number of days next-of-kin is absent from work during the period of sickness of the patient in relation to the admission, number of days next-of-kin is not able to perform daily tasks such as cooking, grocery shopping and house cleaning during the period of sickness of the patient in relation to the admission and number of days in isolation during the period of sickness of the patient in relation to the admission
Organizational related endpoints: Costs of hospital resource use | Three months after discharge of patient
  Economic outcome
Organizational related endpoints: Number of contacts to general practitioner | Three months after discharge of patient
  Economic outcome
Organizational related endpoints: Costs of general practitioner resource use | Three months after discharge of patient
  Economic outcome
Organizational related endpoints: Total costs of health care utilization per patient | Three months after discharge of patient
  Economic outcome
Organizational related endpoints: Intervention costs | Three months after discharge of patient
  Economic outcome
Organizational related endpoints: Number of in-hospital days | Three months after discharge of patient
  Economic outcome
Organizational related endpoints: Number of outpatient visits | Three months after discharge of patient
  Economic outcome
Organizational related endpoints: Productivity losses | Three months after discharge of patient
  Economic outcome: A calculation of the costs in relation to the home admission of the patients during the feasibility study.
Health-related Quality of Life | Three months after discharge of patient
  SF36
Health-related Quality of Life | Three months after discharge of patient
  EQ-5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Thea K Fischer, MD, Principal Investigator — Nordsjaellands Hospital
Locations (1):
- Nordsjaellands Hospital, Hillerød, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sandreva T, Larsen MN, Rasmussen MK, Nielsen TL, von Sydow C, Schmidt TA, Fischer TK. Transforming health care: Investigating Influenzer, a novel telemedicine-supported early discharge program for patients with lower respiratory tract infection: A non-randomized feasibility study. J Telemed Telecare. 2025 Sep;31(8):1138-1151. doi: 10.1177/1357633X241254572. Epub 2024 May 23. PMID 38780386